CLINICAL TRIAL: NCT05033327
Title: The Acceptability of an App-based, Interactive, Personalized Nutrition and Exercise Program to Support Self-management in Cirrhosis: a Pilot Study
Brief Title: Feasibility of an App-based Nutrition & Exercise Program in Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian National Transplant Research Program (Other); Nutricia Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00087451
Record Dates: First submitted 2020-03-23; First posted 2021-09-02 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Cirrhosis, Liver; Hepatic Encephalopathy
MeSH Terms: conditions — Liver Cirrhosis; Hepatic Encephalopathy | interventions — Nutritional Status

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrition and Exercise App (Other): The exercise and nutrition app intervention will be provided to study participants. The app offers self-directed and supervised (virtual) programming to support nutrition and exercise self-management. Each participant follows a program that has been tailored to their overall health, physical function, and needs.
  Interventions: Behavioral: Nutrition and Exercise app

INTERVENTIONS:
Behavioral: Nutrition and Exercise app — Personalized, home-based, interactive therapy app
  Other Names: Heal-Me

SUMMARY:
The personalized nutrition and exercise app was designed for use by individuals living with chronic conditions. The pilot study examines the acceptance and use of the online, interactive program to support self-management in cirrhosis.

DETAILED DESCRIPTION:
Patients living with chronic disease are at-risk for frailty because of their potentially sedentary lifestyle and/or symptoms. Supervised exercise programs are useful for improving or maintaining physical capacity as measured by common physical function measures. However, accessibility is limited due to scheduling, transportation, employment, and residential location. Unsupervised, self-directed home-based programs have had limited success due to absence of peer support and accountability.

An alternative is an app-based program that offers interactive engagement with study staff and accountability. Further, follow-along videos and tracking for both nutrition and exercise can be completed at the patient's convenience.

A 12-week pilot study with patients living with cirrhosis will assess the acceptability of the programming. The hypothesis is that study participants will find the customization of the app and interaction with the study staff acceptable as measured by completion rates (primary study endpoint). Secondary outcomes include change in measures (0-12 weeks) for the 6-minute walk test (6MWT), thigh muscle thickness, and chair sit-to-stands. At the end of the study, participants will also complete a program satisfaction survey (developed in-house).

Interviews with participants, caregivers, and study staff, conducted via videoconference at 4-6 weeks and end of study, will be descriptively analysed to identify feasibility, acceptability, and perceived utility of the program. Analyses will also identify areas for program improvement.

ELIGIBILITY:
Inclusion Criteria:

* adult (aged 18 years and older)
* diagnosis of cirrhosis (MELD<25) according to biopsy, imaging, elastography, or other
* fulfill the guideline-based prophylaxis in place for high risk gastroesophageal varices
* able to communicate (e.g., speak, read, and write) in English
* provide informed written consent for self

Exclusion Criteria:

* hepatocellular carcinoma (HCC) outside of the Edmonton liver transplant criteria
* previous myocardial infarction
* EF <50%
* ischemia on stress testing
* oxygen saturation <95%
* non-HCC malignancy
* end-stage renal disease.
* at the discretion of the healthcare team if a participant can participate in the pilot study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Participant Retention/Adherence | 12 weeks
  The number of participants who complete the 12-week nutrition and exercise program and meet 70% of the nutrition and exercise goals.

SECONDARY OUTCOMES:
6-MWT | 12 weeks
  The change in distance walked in 6 minutes.
Program Satisfaction | 12 weeks
  Self-reported satisfaction with the nutrition and exercise program.

OTHER OUTCOMES:
Chair Sit-to-Stand | 12 weeks
  The change in time required to complete 5x sit-to-stands from baseline to end of study.
Thigh Muscle Measures | 12 weeks
  The change in thigh muscle thickness and echogenicity from baseline to end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Puneeta Tandon, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tandon P, Ismond KP, Riess K, Duarte-Rojo A, Al-Judaibi B, Dunn MA, Holman J, Howes N, Haykowsky MJF, Josbeno DA, McNeely M. Exercise in cirrhosis: Translating evidence and experience to practice. J Hepatol. 2018 Nov;69(5):1164-1177. doi: 10.1016/j.jhep.2018.06.017. Epub 2018 Jun 30. PMID 29964066
- [Background] Eslamparast T, Montano-Loza AJ, Raman M, Tandon P. Sarcopenic obesity in cirrhosis-The confluence of 2 prognostic titans. Liver Int. 2018 Oct;38(10):1706-1717. doi: 10.1111/liv.13876. Epub 2018 May 25. PMID 29738109
- [Background] Mazurak VC, Tandon P, Montano-Loza AJ. Nutrition and the transplant candidate. Liver Transpl. 2017 Nov;23(11):1451-1464. doi: 10.1002/lt.24848. PMID 29072825
- [Background] Ney M, Gramlich L, Mathiesen V, Bailey RJ, Haykowsky M, Ma M, Abraldes JG, Tandon P. Patient-perceived barriers to lifestyle interventions in cirrhosis. Saudi J Gastroenterol. 2017 Mar-Apr;23(2):97-104. doi: 10.4103/1319-3767.203357. PMID 28361840
- [Background] Ney M, Haykowsky MJ, Vandermeer B, Shah A, Ow M, Tandon P. Systematic review: pre- and post-operative prognostic value of cardiopulmonary exercise testing in liver transplant candidates. Aliment Pharmacol Ther. 2016 Oct;44(8):796-806. doi: 10.1111/apt.13771. Epub 2016 Aug 19. PMID 27539029
- [Background] Zenith L, Meena N, Ramadi A, Yavari M, Harvey A, Carbonneau M, Ma M, Abraldes JG, Paterson I, Haykowsky MJ, Tandon P. Eight weeks of exercise training increases aerobic capacity and muscle mass and reduces fatigue in patients with cirrhosis. Clin Gastroenterol Hepatol. 2014 Nov;12(11):1920-6.e2. doi: 10.1016/j.cgh.2014.04.016. Epub 2014 Apr 24. PMID 24768811
- See also: Study website — http://www.wellnesstoolbox.ca